CLINICAL TRIAL: NCT04681339
Title: Antibiotic Prescription in Children Hospitalized for Community-acquired Pneumonia: a Prospective, Observational Study
Brief Title: Antibiotic Prescription in Children Hospitalized for Community-acquired Pneumonia
Status: Recruiting | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Gemeinschaftskrankenhaus Herdecke, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: PKA-03
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Community Acquired Pneumonia in Children; Antibiotic Stewardship
Keywords: Community acquired pneumonia; Antibiotic use; Pediatrics; Hospitalised children; Integrative medicine
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pneumonia with antibiotics: Children with non-severe community acquired pneumonia and fever: managed with antibiotics
  Interventions: Other: Antibiotic treatment
- Pneumonia without antibiotics: Children with non-severe community acquired pneumonia and fever: managed without antibiotics
  Interventions: Other: No antibiotic treatment

INTERVENTIONS:
Other: Antibiotic treatment — Antibiotic treatment
  Groups: Pneumonia with antibiotics
Other: No antibiotic treatment — No antibiotic treatment
  Groups: Pneumonia without antibiotics

SUMMARY:
A study to observe how often antibiotics are prescribed in children hospitalized for pneumonia and how doctors decide if a child needs antibiotics or not. Parent satisfaction will also be recorded.

DETAILED DESCRIPTION:
An observational study to document the antibiotic treatment rate of children hospitalized for community acquired pneumonia at a pediatric department with longstanding practice of restrictive antibiotic prescribing. Patients will be enrolled consecutively and treated according to in-house standard operating procedure. Antibiotic treatment rate, severity of disease and medical complication rate in antibiotic and non-antibiotic managed children, frequency of predefined factors in physician decision making on antibiotic use, and parental satisfaction will be recorded. Parents will be contacted at least 4 weeks after discharge to inquire about recurrence or readmission.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission at the pediatric department of the Filderklinik or at the pediatric department of the Herdecke Community Hospital
* Admission diagnosis pneumonia or pneumonia diagnosis within 48 hours of admission
* Written informed consent by care giver
* All inclusion criteria have to be fulfilled

Exclusion Criteria:

* Insufficient knowledge of German to understand the written patient information and questionnaire

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (aged 3 months to 18 years) who are hospitalized for pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Antibiotic treatment rates in hospitalized children with non-severe community-acquired pneumonia and fever | During hospitalization, an average of 7 days
  Rates of treatment with and without antibiotics during hospitalization

SECONDARY OUTCOMES:
Number of medical complications | During hospitalization, an average of 7 days
  Medical complications defined as a) admission to intensive care, mechanical ventilation, transfer to tertiary car center OR b) pleural effusion or empyema, pneumothorax, lung abscess, bronchopleural fistula, necrotizing pneumonia, acute respiratory failure, infectious complication (meningitis, septic shock).
Factors in physician decision making on antibiotic prescription | During hospitalization, an average of 7 days
  Physician questionnaire (closed-ended questions)
Parental satisfaction | At discharge, assessing the entire duration of the hospital stay, an average of 7 days
  Parental satisfaction questionnaire (closed-ended questions)
Hospitalization duration | At discharge, assessing the entire duration of the hospital stay, an average of 7 days
  Number of hospitalization days
Number of children with relevant comorbidity | During hospitalization, an average of 7 days
  Co-morbidities that may affect decision on antimicrobial use: a) chronic conditions (e.g. neurological conditions such as cerebral palsy, Down syndrome; or chronic respiratory conditions such as asthma, cystic fibrosis; or heart conditions). b) acute infectious comorbidities: bronchiolitis, otitis media, urinary tract infection, confirmed influenza virus or Respiratory Syncytial Virus or SARS-CoV2.
Days of supplemental oxygen use | During hospitalization, an average of 7 days
  Oxygen therapy for O2 saturation <92%
Use of antipyretic medications | During hospitalization, an average of 7 days
  Number of doses of paracetamol or ibuprofen during hospitalization
Number of complementary medicine medications used per child | During hospitalization, an average of 7 days
  Number of complementary medication during hospitalization
Number of readmissions for pneumonia or new pneumonia recurrences within 4 weeks of hospital discharge | 4 weeks after end of hospitalization
  New hospital admission for pneumonia; treatment requiring recurrence of pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr, Principal Investigator — Arcim Institute
Locations (2):
- Germany (2):
  - Die Filderklinik, Filderstadt, Baden-Wurttemberg
  - Herdecke Community Hospital, Herdecke, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.